CLINICAL TRIAL: NCT05766943
Title: The Efficacy of the Smart Pass Filter to Reduce the Risk for Inappropriate Subcutaneous Implantable Cardioverter-defibrillator Shocks From Myopotential Interference
Brief Title: Reduction of Myopotential Interference With Smart Pass in S-ICD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Michael Gold, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 00117025
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Subcutaneous ICD; Myopotential Interference
Keywords: Device interrogation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Smart Pass ON (Active Comparator): Smart Pass filter will be programmed ON in the S-ICD while performing exercise testing.
  Interventions: Device: Smart Pass ON
- Smart Pass OFF (Placebo Comparator): Smart Pass filter will be programmed OFF in the S-ICD while performing exercise testing.
  Interventions: Device: Smart Pass OFF

INTERVENTIONS:
Device: Smart Pass ON — Smart Pass filter will be programmed ON in the S-ICD while performing exercise testing.
  Arms: Smart Pass ON
Device: Smart Pass OFF — Smart Pass filter will be programmed OFF in the S-ICD while performing exercise testing.
  Arms: Smart Pass OFF

SUMMARY:
This study is enrolling participants who are already implanted with a S-ICD device ( subcutaneous ICD), and are undergoing a routine outpatient clinic follow up appointment to have their S-ICD checked. The aim of the study is to see if a feature in the device can recognize muscle movement and differentiate movement from irregular heart signals. The study involves doing some simple arm exercises while collecting device data, both with this feature turn on and then with it turned off. Participants will be randomized to either have the feature turned on or off initially then it will be programmed the alternative way and the same exercise testing will be repeated. The study will involve just one visit.

DETAILED DESCRIPTION:
This study is enrolling participants who are already implanted with a S-ICD device ( subcutaneous ICD), and are undergoing a routine outpatient clinic follow up appointment to have their S-ICD checked. The aim of the study is to see if a feature in the device can recognize muscle movement and differentiate movement from irregular heart signals. The study involves doing some simple arm exercises while collecting device data, both with this feature turn on and then with it turned off. Participants will be randomized to either have the feature turned on or off initially, then it will be programmed the alternative way and the same exercise testing will be repeated. The study will involve just one visit. Following this visit study participation is complete.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Implanted EMBLEM S-ICD (Model A 209 and Model A 219, Boston Scientific, St Paul, MN, USA)

Exclusion Criteria:

* Less than 18 years of age
* Hemodynamically unstable
* Inability to preform TET due to orthopedic issues or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of myopotential interference | throughout the intervention, approximately 20 minutes
  The incidence of myopotential interference, assessed by subcutaneous electrogram annotated "T" marker during the tube exercise test with or without Smart Pass filter

SECONDARY OUTCOMES:
Incidence of MPI in US participants and Japanese participants | duration of enrollment, approximately 6 months
  Compare the differences in the incidence of myopotential interference in US and Japanese participants

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Gold, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No